CLINICAL TRIAL: NCT02964572
Title: Effect of Sodium Glucose Co-transporter 2 Inhibitor on Inflammatory Cytokine in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0795
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — glimepiride; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride (Active Comparator): Glimepiride (anti-diabetic drug) as a comparison group
  Interventions: Drug: Glimepiride
- Empagliflozin (Experimental): Empagliflozin (anti-diabetic drug) as a study group
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Glimepiride — In accordance with the standard treatment guidelines of diabetes, glimepiride as a drug of active comparator will be administered to improve blood sugar in patients with poorly controlled blood sugar.
  Other Names: Amaryl
  Arms: Glimepiride
Drug: Empagliflozin — Empagliflozin as a drug of experimental will be administered to improve blood sugar in patients with poorly controlled blood sugar.
  Other Names: Jardiance
  Arms: Empagliflozin

SUMMARY:
* Single-center, prospective, active-controlled, open, randomized, 2 arm parallel, interventional, exploratory pilot
* Type 2 diabetic patients with high cardiovascular risks who have inadequate glycaemic control with metformin-based oral hypoglycemic agents will be prescribed glimepiride (comparison group) or empagliflozin (study group) for 60 days (plus or minus 32 days) as add-on therapy
* Changes in IL-1beta secretion, serum beta-hydroxybutyrate concentration, and NLRP3 inflammasome activity from baseline to final timepoint will be assessed.

DETAILED DESCRIPTION:
First among cardiovascular (CV) end point trials of glucose-lowering agents, the EMPA-REG OUTCOME trial-using 10 or 25 mg/day SGLT2 inhibitor empagliflozin against placebo in 7,020 patients with T2DM who were at increased CV risk-reported a 14% reduction in major CV events and marked relative risk reductions in CV mortality (38%), hospitalization for heart failure (35%), and death from any cause (32%) over a median time period of 2.6 years. Though these results have raised the possibility that mechanisms other than those observed in the trial-modest improvement in glycemic control, small decrease in body weight, and persistent reductions in blood pressure and uric acid level-may be at play, it's not clearly known yet.

The inflammatory nature of atherosclerosis is well established. We hypothesized that empagliflozin might have an inhibitory effect on inflammasome activity in macrophages, thus contribute to cardioprotective effects in diabetes.

* Single-center, prospective, active-controlled, open, randomized, 2 arm parallel, interventional, exploratory pilot
* Type 2 diabetic patients with high cardiovascular risks who have inadequate glycaemic control with metformin-based oral hypoglycemic agents will be prescribed glimepiride (comparison group) or empagliflozin (study group) for 60 days (plus or minus 32 days) as add-on therapy
* Changes in IL-1beta secretion, serum beta-hydroxybutyrate concentration, and NLRP3 inflammasome activity from baseline to final timepoint will be assessed
* Healthy volunteers : effect of 3 day-ketogenic diet on changes in cytokines, metabolites (IL-1beta, beta-hydroxybutyrate , etc) and inflammasome activity in macrophages

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years
* inadequate glycaemic control : HbA1c ≥6.5% or fasting glucose >120 mg/dl or random glucose >180 mg/dl
* High risk of cardiovascular events defined as the presence of ≥1 of the following:

  1. History of myocardial infarction
  2. Evidence of multi-vessel coronary artery disease
  3. Evidence of single-vessel coronary artery disease with a positive non-invasive stress test for ischemia or history of hospitalization for unstable angina
  4. History of stroke
  5. Evidence of occlusive peripheral artery disease
  6. Evidence of carotid atherosclerosis
  7. Metabolic syndrome
* Healthy volunteers

Exclusion Criteria:

* Type 1 diabetes
* Organ transplantation
* Pregnant women
* eGFR <45
* Cortisol or growth hormone deficiency, pituitary diseases
* Gastric surgery
* Hematologic disorders
* Active cancers

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
changes in the secretion of IL-1 beta from peripheral blood mononuclear cells | Day 60
  The effect of empagliflozin on the secretion of IL-1beta from peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Changes in the secretion of TNF-alpha from peripheral blood mononuclear cells, before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of beta-hydroxybutyrate, before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in body weight (kg), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of insulin (µU/mL), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of glucagon (pg/mL), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of free fatty acid (μEq/L), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum glycated albumin (%), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of glucose (mg/dL), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of uric acid (mg/dL), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of liver enzymes (aspartate aminotransferase and alanine aminotransferase (IU/L)), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum lipids (total cholesterol, triglyceride, HDL cholesterol, and LDL cholesterol (mg/dL)), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in serum concentrations of creatinine (mg/dL), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in spot urine concentrations of glucose (mg/dL) and creatinine (mg/dL) (those will be combined to report spot urine glucose-to-creatinine ratio in mg/mg), before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in mRNA expression level (PCR, fold) of IL-1beta, TNF-alpha, and NLRP3 in peripheral blood mononuclear cells, before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days
Changes in protein expression pattern (western blot, relative to control) of IL-1beta, TNF-alpha, and NLRP3 in peripheral blood mononuclear cells, before and after the administration of empagliflozin or glimepiride | Day 60 plus or minus 32 days

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of Internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim ER, Kim SR, Cho W, Lee SG, Kim SH, Kim JH, Choi E, Kim JH, Yu JW, Lee BW, Kang ES, Cha BS, Lee MS, Cho JW, Jeon JY, Lee YH. Short Term Isocaloric Ketogenic Diet Modulates NLRP3 Inflammasome Via B-hydroxybutyrate and Fibroblast Growth Factor 21. Front Immunol. 2022 Apr 28;13:843520. doi: 10.3389/fimmu.2022.843520. eCollection 2022. PMID 35572519